CLINICAL TRIAL: NCT07180160
Title: Iparomlimab and Tuvonralimab (QL1706) in Patients With Hormone Receptor-positive, Human Epidermal Growth Factor Receptor 2-negative Advanced Breast Cancer: a Prospective, Randomised, Controlled, Multicentre Clinical Trial
Brief Title: Iparomlimab and Tuvonralimab (QL1706) in Patients With HR-positive, HER2-negative Advanced Breast Cancer
Acronym: ITHRAN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wenjin Yin (Other)
Responsible Party: Sponsor-Investigator, Wenjin Yin, Deputy Chief of Breast Surgery Department, RenJi Hospital
Organization: RenJi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY2025-215-C
Record Dates: First submitted 2025-09-10; First posted 2025-09-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1706 (Experimental): QL1706 + CDK4/6 inhibitor + fulvestrant/letrozole
  Interventions: Drug: QL1706; Drug: CDK4/6 inhibitor; Drug: Fulvestrant
- control (Active Comparator): CDK4/6 inhibitor + fulvestrant/letrozole
  Interventions: Drug: CDK4/6 inhibitor; Drug: Fulvestrant

INTERVENTIONS:
Drug: QL1706 — QL1706 is a single bifunctional MabPair product consisting of two engineered monoclonal antibodies (anti-PD-1 and anti-CTLA-4).
  Arms: QL1706
Drug: CDK4/6 inhibitor — palbociclib OR ribociclib OR abemaciclib OR dalpiciclib
Drug: Fulvestrant — SERD

SUMMARY:
This is a prospective, randomised, controlled, multicentre study to evaluate the efficacy and safety of Iparomlimab and Tuvonralimab (QL1706) in patients with hormone receptor-positive/human epidermal growth factor receptor 2-negative advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female, age≥18 years old
* Expected survival ≥12 weeks
* ECOG 0-1
* Pathologically confirmed recurrent or metastatic breast cancer not amenable to curative surgery
* ER and/or PR positive, HER2 negative
* At least one measurable lesion or bone-only disease (osteolytic or mixed) according to RECIST v1.1
* Previously treated with ≤2 lines chemotherapy for advanced disease; previously treated with ≤2 CDK4/6 inhibitors
* Adequate organ function

Exclusion Criteria:

* During pregnancy and lactation
* Patients with central nervous system metastasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the date of starting study treatment to the date of first documentation of disease progression or death from any cause (up to approximately 1 year)
  PFS is defined as the time from the date of starting maintenance therapy to the date of disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Adverse events | From the date of starting study treatment to the end of the treatment (up to approximately 1 year)
  Adverse events during maintenance therapy will be assessed according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjin Yin, M.D., Principal Investigator — Renji Hospital,School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No